CLINICAL TRIAL: NCT03701854
Title: Comparison of Functional and Maximal Exercise Capacity, Respiratory and Peripheral Muscle Strength, Dyspnea and Fatigue in Heart Failure Patients With Pacemakers and Healthy Controls
Brief Title: Physical Impairments in Heart Failure Patients With Pacemakers
Status: Completed | Type: Observational
Sponsor: Gazi University (Other)
Responsible Party: Principal Investigator, Meral Boşnak Güçlü, Associate professor, Gazi University
Other Study IDs: GaziUniversity16
Record Dates: First submitted 2018-10-05; First posted 2018-10-10 (Actual); Last update posted 2018-10-10 (Actual); Status verified 2018-10

CONDITIONS: Heart Failure Patients
Keywords: heart failure; pacemaker; exercise test; muscle strength; dyspnea; fatigue
MeSH Terms: conditions — Heart Failure; Dyspnea; Fatigue

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Heart failure patients with pacemakers: Functional (6-Minute Walking test (6-MWT)) and maximal exercise capacity (Incremental Shuttle Walking test (ISWT)), respiratory (MIP, MEP; Mouth pressure device) and peripheral muscle strength (Dynamometer), pulmonary function (Spirometry) dyspnea (Modified Medical Research Council Dyspnea scale) (MMRC)), and fatigue (Fatigue Severity scale (FSS)) were evaluated in 50 patients.
- Healthy controls: Healthy individuals (n=40) were selected from individuals without known and diagnosed any chronic diseases. Similar measurements were applicated in healthy individuals.

SUMMARY:
Despite major breakthroughs that have recently been made in pacemakers implanted in heart failure (HF) patients, it is clear that functional impairments and symptoms often remain. However, only limited studies have investigated exercise capacity, muscle strength, pulmonary function, dyspnea, and fatigue in pacemaker implanted HF patients. Therefore, investigators aimed to compare the aforementioned outcomes in patients and healthy controls.

DETAILED DESCRIPTION:
Heart failure is a chronic, progressive condition in which the heart muscle is unable to pump enough blood through to meet the body's needs for blood and oxygen. Safeguarding HF patients at increased risk of sudden cardiac death due to ventricular arrhythmias and HF as a result of left ventricular systolic dysfunction and cardiac abnormal synchronization has continued to improve. Implantable cardioverter defibrillators (ICDs), which restore normal heart rhythm using pacing, cardioversion or defibrillation, and cardiac resynchronization therapy (CRT), which resynchronizes the contraction of the heart using biventricular pacing, are nowadays widely used to treat the aforementioned conditions.

New developments in medical treatments have focused on the primary affected organs, targeting reduced left ventricular ejection fraction in chronic HF. Although major breakthroughs in the treatments have occurred in recent years, especially implantable medical devices, it is clear that when drugs are optimally prescribed, even the latest technology used in pacemakers reported problems, especially functional impairments and symptoms often remain. In recent decades, it has become obvious that disease severity should not be estimated from cardiac function impairment alone. However, what has not hitherto been clearly investigated is the fact that even functional and maximal exercise capacity, respiratory and peripheral muscle strength and pulmonary function are impaired, and dyspnea in the activities of daily living and fatigue perception increased in HF patients with pacemakers.

Hence, investiators designed a prospective, cross-sectional study to compare the aforementioned outcomes in HF patients with pacemakers and healthy controls. Investigators hypothesized that functional and maximal exercise capacity, respiratory and peripheral muscle strength, and pulmonary function are impaired, and dyspnea in the activities of daily living, and fatigue perception increased in HF patients with pacemakers.

A cross-sectional study. 50 HF patients with pacemakers and 40 controls were compared. Functional (6-Minute Walking test (6-MWT)) and maximal exercise capacity (Incremental Shuttle Walking test (ISWT)), respiratory (MIP, MEP; Mouth pressure device) and peripheral muscle strength (Dynamometer), pulmonary function (Spirometry) dyspnea (Modified Medical Research Council Dyspnea scale) (MMRC)), and fatigue (Fatigue Severity scale (FSS)) were evaluated.

ELIGIBILITY:
Inclusion criteria:

* Heart failure patients with ischemic or non-ischemic etiology,
* Aged between 18 and 80 years,
* Being clinically stable for at least 4 weeks,
* Having any type of implantable cardioverter-defibrillator (ICD), cardiac resynchronization therapy (CRT), New York Heart Association (NYHA) Class II-III,
* Having no change in medications over three months and all comorbid conditions, such as hypertension and diabetes, controlled.

Exclusion criteria:

* Having acute myocardial infarction, cognitive disorders, complex arrhythmias, uncontrolled hypertension, stroke or transient ischemic attack within the last six months prior to the study, angina pectoris, recent viral infections (six months prior to study), significant valvular disease,
* Having history of malignancy,
* Having orthopedic problems and rheumatologic diseases.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Prior to evaluation, all patients' clinical evaluation and echocardiographic measurements and pacemaker routine controls were conducted by a cardiologist. All patients and controls were tested by a physical therapist. Demographic characteristics were recorded. Functional and maximal exercise capacity, respiratory and peripheral muscle strength, pulmonary function, dyspnea and fatigue perception were evaluated and compared with age- and gender-matched healthy controls (without any chronic diseases) who volunteered to participate to the study.
Sampling Method: Non-Probability Sample
Enrollment: 138 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2018-08-30 (Actual); Study Completion 2018-08-30 (Actual)

PRIMARY OUTCOMES:
submaximal exercise capacity evaluation | 8-10 minutes
  The six-minute walking test (6-MWT) was used to evaluate submaximal exercise capacity.

SECONDARY OUTCOMES:
pulmonary function test | 5 minutes
  This test was evaluated using a spirometry by which is evaluated dynamic lung functions expressed as percentages of expected values.
inspiratory and expiratory muscle strength (MIP, MEP) | 5-10 minutes
  Respiratory muscle strength was evaluated with a mouth pressure device
peripheral muscle strength | 10 minutes
  Peripheral muscle strength was evaluated with a hand-held dynamometer
fatigue severity | 1-3 minutes
  The Turkish version of Fatigue Severity Scale, which is a valid and reliable test, was performed to the recipients for evaluation of fatigue severity. Self-administered questionnaire is comprised of nine questions. The average score is identified on seven-point scale. Patients select a number from 1 to 7 for each 9 questions which demonstrates from strong disagreement to strong agreement, respectively. The cut-off score for fatigue severity is 36 according to this scale, if the total score obtained from this scale is higher than 36, the recipient is defined as severe fatigue.
Dyspnea severity | 2 minutes
  The severity of dyspnea during daily living activities was evaluated using the Modified Medical Research Council (MMRC) dyspnea scale. Dyspnea is graded as follows: zero (dyspnea only with strenuous exercise), one (dyspnea when hurrying or walking up a slight hill), two (walks slower than people of the same age due to dyspnea or having to stop for breath when walking at own pace), three (stops for breath after walking 100 yards or after a few minutes) and four (too dyspneic to leave house or breathless when dressing). The minimal clinically important difference (MCID) is 1 unit for the MMRC dyspnea scale.
maximal exercise capacity evaluation | 10-15 minutes
  and the incremental shuttle walk test (ISWT) was used to evaluate submaximal exercise capacity.

CONTACTS AND LOCATIONS:
Overall Officials: Meral Boşnak Güçlü, PhD, Study Director — Gazi University; Gülşah Barğı, PhD, Study Chair — Gazi University; Nihan Katayıfçı, MsC, Study Chair — Mustafa Kemal Üniversitesi Fizik Tedavi ve Rehabilitasyon Yüksekokulu Fizyoterapi ve Rehabilitasyon Bölümü; Fatih Şen, PhD., Study Chair — Mustafa Kemal Üniversitesi Tayfur Ata Sökmen Tıp Fakültesi Kardiyoloji Anabilim Dalı
Locations (1):
- Gazi University Faculty of Health Science Department of PhysioTherapy, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
There is not a plan to make individual participant data but when the statistical analyses of all data are made, all results will be shared.

REFERENCES:
- [Background] Jonsdottir S, Andersen KK, Sigurosson AF, Sigurosson SB. The effect of physical training in chronic heart failure. Eur J Heart Fail. 2006 Jan;8(1):97-101. doi: 10.1016/j.ejheart.2005.05.002. Epub 2005 Sep 27. PMID 16194620
- [Background] Clark AL. Origin of symptoms in chronic heart failure. Heart. 2006 Jan;92(1):12-6. doi: 10.1136/hrt.2005.066886. Epub 2005 Sep 13. PMID 16159969
- [Background] Volterrani M, Clark AL, Ludman PF, Swan JW, Adamopoulos S, Piepoli M, Coats AJ. Predictors of exercise capacity in chronic heart failure. Eur Heart J. 1994 Jun;15(6):801-9. doi: 10.1093/oxfordjournals.eurheartj.a060588. PMID 8088269
- [Background] Buller NP, Jones D, Poole-Wilson PA. Direct measurement of skeletal muscle fatigue in patients with chronic heart failure. Br Heart J. 1991 Jan;65(1):20-4. doi: 10.1136/hrt.65.1.20. PMID 1993126
- [Background] Minotti JR, Pillay P, Chang L, Wells L, Massie BM. Neurophysiological assessment of skeletal muscle fatigue in patients with congestive heart failure. Circulation. 1992 Sep;86(3):903-8. doi: 10.1161/01.cir.86.3.903. PMID 1516203